CLINICAL TRIAL: NCT05265923
Title: A Randomized, Double Blind, Placebo-controlled Phase 3 Study to Evaluate the Efficacy and Safety of CM310 in Patients With Moderate-to-severe Atopic Dermatitis
Brief Title: A Study of CM310 in Patients With Moderate-to-Severe Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM310AD005
Record Dates: First submitted 2022-02-17; First posted 2022-03-04 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CM310 (Experimental): CM310, 600mg for the initial dose, and 300mg for subsequent doses, subcutaneous injection (SC), every 2 weeks (Q2W)
  Interventions: Drug: CM310
- Placebo (Placebo Comparator): Double blind treatment period : Placebo
  Maintenance treatment period : CM310, 600mg for the initial dose, and 300mg for subsequent doses, subcutaneous injection (SC), every 2 weeks (Q2W)
  Interventions: Drug: CM310; Other: Placebo

INTERVENTIONS:
Drug: CM310 — IL-4Rα monoclonal antibody
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double blind, placebo-controlled phase 3 study to evaluate the efficacy, safety, PK, PD and immunogenicity of CM310 in patients with moderate-to-severe atopic dermatitis.

DETAILED DESCRIPTION:
The study consists of an up-to-4-week screening period, a 16-week double-blind treatment period, a 36-week maintenance treatment period, and a 8-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with AD for at least 12 months before Screening, with below requirements: 1) EASI score ≥16 at Screening and Baseline; 2) IGA score ≥3 at Screening and Baseline; 3) ≥10% BSA of AD involvement at Screening and Baseline; 4) Pruritus NRS average score ≥3 at Baseline.

Exclusion Criteria:

* Not enough washing-out period for previous therapy.
* Concurrent disease/status which may potentially affect the efficacy/safety judgement.
* Organ dysfunction.
* pregnancy.
* Other.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving EASI-75 at week 16 | 16 weeks
  Proportion of subjects achieving EASI-75 (≥75% reduction from baseline in Eczema Area and Severity Index score) at week 16.
  The EASI is a composite index with scores ranging from 0 to 72. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) will each be assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe).
Proportion of subjects with IGA score of 0 or 1 and a reduction of IGA score by ≥2 points from baseline at week 16 | 16 weeks
  Proportion of subjects with Investigator's Global Assessment (IGA) score of 0 or 1 and a reduction of IGA score by ≥2 points from baseline at week 16.
  IGA is an assessment instrument used in clinical studies to rate the severity of AD globally, based on a 5-point scale ranging from 0 (clear) to 4 (severe).

SECONDARY OUTCOMES:
Incidence of adverse events (AEs), abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing. | 64 weeks
  Incidence of adverse events (AEs), abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing.
Percent change of EASI score from baseline | 52 weeks
  The EASI is a composite index with scores ranging from 0 to 72. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) will each be assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe).
Percent change of NRS score from baseline | 52 weeks
  The range of Pruritus Numerical Rating Scale (NRS) is from 0 (no itch)-10 (worst imaginable itch)
Body surface area (BSA) of involvement of atopic dermatitis | 52 weeks
  Change from baseline in percent of BSA
Changes from baseline in Dermatology Life Quality Index (DLQI) | 52 weeks
  The DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on quality of life. It is a 10-question questionnaire with a score of 0 (not at all) to 3 (very much) for each question. A high score is indicative of a poor quality of life.
Immunogenicity: anti-drug antibody (ADA) and neutralizing antibody (Nab) | 64 weeks
  anti-drug antibody (ADA) and neutralizing antibody (Nab)

CONTACTS AND LOCATIONS:
Overall Officials: jianzhong zhang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's hospital, Beijing, China

REFERENCES:
- [Derived] Zhao Y, Zhang L, Wu L, Yang B, Wang J, Li Y, Diao Q, Li J, Sun Q, Zhu X, Man X, Wang L, Feng Y, Cai T, Zeng H, Li L, Lu J, Ren H, Li F, Lu Q, Tao X, Xiao R, Ji C, Zhao W, Chu W, Chen B, Zhang J. Efficacy and Safety of Stapokibart in Adults With Moderate-to-Severe Atopic Dermatitis With and Without Type 2 Comorbidities: A Post Hoc Analysis of a Phase 3 Trial. Clin Transl Allergy. 2025 Nov;15(11):e70121. doi: 10.1002/clt2.70121. PMID 41257453
- [Derived] Zhao Y, Zhang L, Wu L, Yang B, Wang J, Li Y, Diao Q, Li J, Sun Q, Zhu X, Man X, Wang L, Feng Y, Cai T, Zeng H, Li L, Lu J, Ren H, Li F, Lu Q, Tao X, Xiao R, Ji C, Liang C, Qiu Y, Chen B, Zhang J. Patient-Reported Outcomes in Adults with Moderate-to-Severe Atopic Dermatitis Treated with Stapokibart over 52 weeks: A Post Hoc Analysis of a Phase 3 Trial. Adv Ther. 2025 Sep;42(9):4527-4539. doi: 10.1007/s12325-025-03284-7. Epub 2025 Jul 12. PMID 40650707